CLINICAL TRIAL: NCT01498848
Title: Effect of Cooking Oils on Whole Blood and Saliva Fatty Acids in Children in Bogota, Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, ANA BAYLIN, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00048757
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soybean oil (Active Comparator): Families were given soybean oil for cooking during 4 weeks
  Interventions: Dietary Supplement: Cooking oils
- Sunflower oil (Active Comparator): Families were given sunflower oil for cooking during 4 weeks
  Interventions: Dietary Supplement: Cooking oils

INTERVENTIONS:
Dietary Supplement: Cooking oils — Families were randomized to receive either soybean or sunflower oil for cooking during 4 weeks

SUMMARY:
We conducted a randomized trial to determine the effect of providing families from Bogota, Colombia, with a one month supply of one of two cooking oils, sunflower oil vs. soybean oil, on whole blood and saliva fatty acid composition of children. The aims were: 1) assess the effect of the oils on whole blood fatty acid composition in children, 2) assess the correlation between whole blood and saliva to evaluate if fatty acids measured in saliva would be adequate biomarkers of intake. The study was conducted in the context of an ongoing cohort study of school children from Bogotá, Colombia (HUM00043252). We conducted an intervention trial of 4 week duration. Participant families were randomly assigned to either sunflower oil or soybean oil. Families were visited two times during the 4 week period. We collected dietary information from the person in the household in charge of food preparation, and from the child. At the end of the intervention we collected information on whether or not they liked the oil and whether they would be willing to use it, exclusively, for two years, to assess acceptability for a longer intervention. We also collected two finger prick blood samples and two saliva/cheek cells samples from the child, at the beginning and at the end of the study, to evaluate compliance and to assess the impact of the intervention.

DETAILED DESCRIPTION:
We conducted a randomized trial to determine the effect of providing families from Bogota, Colombia, with a one month supply of one of two cooking oils, sunflower oil vs. soybean oil, on whole blood and saliva fatty acid composition of children. The aims were: 1) assess the effect of the oils on whole blood fatty acid composition in children, 2) assess the correlation between whole blood and saliva to evaluate if fatty acids measured in saliva would be adequate biomarkers of intake. The study was conducted in the context of an ongoing cohort study of school children from Bogotá, Colombia (HUM00043252). We conducted an intervention trial of 4 week duration. Participant families were randomly assigned to either sunflower oil or soybean oil. Families were visited two times during the 4 week period. We collected dietary information from the person in the household in charge of food preparation, and from the child. At the end of the intervention we collected information on whether or not they liked the oil and whether they would be willing to use it, exclusively, for two years, to assess acceptability for a longer intervention. We also collected two finger prick blood samples and two saliva/cheek cells samples from the child, at the beginning and at the end of the study, to evaluate compliance and to assess the impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being a participant in the ongoing Bogota School Children cohort

Exclusion Criteria:

* None

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Effect of the intervention on whole blood and saliva fatty acid composition | 4 weeks
  We measured fatty acids in blood to assess effectiveness of the intervention. We measured fatty acids in saliva to evaluate if they can be good biomarkers of intake.

SECONDARY OUTCOMES:
Acceptability and Blindness | 4 weeks
  We assessed acceptability and blindness of the cooking oil intervention by use of questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ana Baylin, MD, DrPH, Principal Investigator — University of Michigan
Locations (1):
- Universidad Pontificia Javeriana, Bogotá, Colombia